CLINICAL TRIAL: NCT00586820
Title: Role of Endothelin in Microvascular Dysfunction Following Percutaneous Coronary Intervention for Non-ST Elevation Myocardial Infarction
Brief Title: Role of Endothelin in Microvascular Dysfunction Following PCI for NSTEMI
Acronym: BQ-123
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amir Lerman, Professor of Medicine, College of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 859-05
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Results first posted 2014-07-04 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-06

CONDITIONS: Myocardial Reperfusion Injury
Keywords: Coronary Atherosclerosis; Microvascular Dysfunction; Non-ST Elevation Myocardial Infarction
MeSH Terms: conditions — Myocardial Reperfusion Injury; Coronary Artery Disease; Non-ST Elevated Myocardial Infarction | interventions — cyclo(Trp-Asp-Pro-Val-Leu)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BQ-123 (Experimental): BQ-123 will be infused at 300 nmol/min for 20 minutes prior to percutaneous coronary intervention (PCI).
  Interventions: Drug: BQ-123
- Placebo (Placebo Comparator): Subjects randomized to the placebo arm will receive a placebo infusion (saline) for 20 minutes prior to PCI.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BQ-123 — BQ-123 is a cyclic peptide consisting of five amino acids. BQ-123 will be infused at 300 nmol/min for 20 minutes prior to percutaneous coronary intervention (PCI).
  Arms: BQ-123
Drug: Placebo — Subjects randomized to the placebo arm will receive a placebo infusion (saline) for 20 minutes prior to PCI.
  Arms: Placebo

SUMMARY:
Percutaneous coronary intervention (PCI) for acute coronary syndromes frequently fails to restore myocardial perfusion despite establishing epicardial vessel patency. Endothelin-1 (ET-1) is a potent vasoconstrictor and its expression is increased in atherosclerotic coronary arteries. Our hypothesis is that increased activity of the endogenous endothelin system contributes to microvascular dysfunction, and adjunctive therapy with an endothelin receptor antagonist will result in improved microvascular blood flow.

Aims: The aims of the study are to assess in patients with non ST-elevation myocardial infarction, whether: 1) PCI causes an increase in coronary blood ET-1 level; 2) an endothelin receptor antagonist acutely improves coronary microvascular blood flow following PCI.

Non-ST segment elevation myocardial infarction (NSTEMI) is one type of heart attack. It is defined as the development of heart muscle necrosis results from an acute interruption of blood supply to a part of the heart which is demonstrated by an elevation of cardiac markers Creatinine Kinase Isoenzyme Muscle/Brain Type (CK-MB) in the blood and the absence of ST-segment elevation in ECG (electrocardiography). ST-segment is a portion of ECG, its elevation indicates full thickness damage of heart muscle. Absence of ST-segment elevation in NSTEMI indicates partial thickness damage of heart muscle occurs. Therefore, NSTEMI is less severe type of heart attack compared to STEMI (ST-segment elevation myocardial infarction) in which full thickness damage of heart muscle occurs.

DETAILED DESCRIPTION:
Our hypothesis is that the endogenous endothelin system contributes to microvascular dysfunction and impaired myocardial reperfusion following successful PCI for non ST-elevation MI, and that endothelin receptor antagonism will improve microvascular flow. The study will provide new insight into the humoral regulation of the microcirculation in patients presenting with acute coronary syndromes.

General methods: This section describes our approach to investigating the specific aims. The study is a prospective, double blind, placebo-controlled trial to assess the efficacy of a selective endothelin type A receptor antagonist (BQ-123), as adjunctive therapy for PCI for non ST elevation MI. The control group will receive placebo rather than another vasodilator in order to specifically elucidate the role of the endogenous endothelin system.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical diagnosis of unstable angina or non ST-elevation myocardial infarction, and requiring clinically indicated PCI for the management of non ST elevation acute coronary syndrome.

Exclusion Criteria:

* Systemic hypotension (systolic <90 mmHg)
* Heart failure or known ejection fraction < 30%
* Left main disease
* Culprit lesion is in a saphenous vein graft
* 100% occlusion of the culprit vessel or culprit is an ostial right coronary stenosis
* Currently enrolled in other active cardiovascular investigational studies
* Severe endocrine, hepatic, or renal disorders
* Pregnancy or lactation
* Federal Medical Center inmates
* Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhiram Prasad, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Guddeti RR, Prasad A, Matsuzawa Y, Aoki T, Rihal C, Holmes D, Best P, Lennon RJ, Lerman LO, Lerman A. Role of endothelin in microvascular dysfunction following percutaneous coronary intervention for non-ST elevation acute coronary syndromes: a single-centre randomised controlled trial. Open Heart. 2016 Aug 4;3(2):e000428. doi: 10.1136/openhrt-2016-000428. eCollection 2016. PMID 27547429

RESULTS

PARTICIPANT FLOW:
Groups:
- BQ-123: The selective endothelin type A receptor antagonist (BQ-123) will be infused at 300 nmol/min for 20 minutes prior to percutaneous coronary intervention (PCI).
Period: Overall Study
Arm/Group | BQ-123 | Placebo
Started | 12 | 11
Completed | 11 | 11
Not Completed | 1 | 0
Not completed — Unsuccessful PCI | 1 | 0

BASELINE CHARACTERISTICS:
Population: 12 subjects were enrolled on the BQ-123 arm, but 1 subject was excluded due to unsuccessful PCI.
Groups:
- Total: Total of all reporting groups
Arm/Group | BQ-123 | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (11.2) | 64 (12.5) | 64.27 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Average Peak Velocity (APV) Immediately Following Percutaneous Coronary Intervention (PCI)
Description: Coronary microvascular blood flow will be assessed following successful PCI by measuring APV in the culprit vessel using Doppler echocardiography.
Time Frame: immediately following PCI procedure
Population: One subject on the BQ-123 arm was excluded from the analysis due to unsuccessful PCI.
Measure: Median (Inter-Quartile Range); unit: cm/s
Arm/Group | BQ-123 | Placebo
Number analyzed (Participants) | 11 | 11
cm/s | 30 [20 to 37] | 19 [9 to 26]
Statistical Analysis 1: Comparison: BQ-123 vs Placebo; Test type: Superiority or Other; p = 0.029, t-test, 2 sided

2. Secondary Outcome: Percent Change in Creatinine Kinase Isoenzyme Muscle/Brain Type (CK-MB) From Immediately Pre-PCI to 8 and 16 Hours Post-PCI
Description: CK-MB is a cardiac marker that can demonstrate the development of heart muscle necrosis resulting from an acute interruption of blood supply to a part of the heart. CK-MB is measured by a blood test.
Time Frame: immediately pre-PCI, 8 hours post-PCI, 16 hours post-PCI
Population: One subject on the BQ-123 arm was excluded from the analysis due to unsuccessful PCI.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | BQ-123 | Placebo
Number analyzed (Participants) | 11 | 11
percent change
  % Change immediate pre-PCI, 8 hr post-PCI | -17 [-26 to -10] | 26 [-15 to 134]
  % Change immediate pre-PCI, 16 hr post-PCI | -17 [-38 to 14] | 107 [2 to 446]
Statistical Analysis 1: Comparison: BQ-123 vs Placebo; Change between the groups from immediate pre-PCI and 8 hours post PCI; Test type: Superiority or Other; p = 0.019, t-test, 2 sided
Statistical Analysis 2: Comparison: BQ-123 vs Placebo; Change between the groups from immediate pre-PCI and 16 hours post-PCI; Test type: Superiority or Other; p = 0.007, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Placebo: Subjects randomized to the placebo arm will receive a placebo infusion for 20 minutes prior to PCI.
Arm/Group | BQ-123 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No